CLINICAL TRIAL: NCT00182559
Title: The Vienna Prograf and Endothelial Progenitor Cell Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gere Sunder-Plassmann, Principal Investigator Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2004-004209-98; 393/2004 (Other: Ethics Committee Medical University of Vienna)
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: End Stage Renal Disease
Keywords: kidney; transplantation; tacrolimus; cyclosporine; conversion
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Cyclosporine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ciclosporin (Active Comparator): Maintain ciclosporin in combination with/without mycophenolate mofetil and with/without steroids at target trough levels of 70-150ng/mL.
  Interventions: Drug: Ciclosporin
- Tacrolimus (Active Comparator): Conversion from ciclosporin to tacrolimus at target trough levels of 5-8 ng/mL in combination with/without mycophenolate mofetil and with/without steroids.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Ciclosporin — Maintain ciclosporin in combination with/without mycophenolate mofetil and with/without steroids at target trough levels of 70-150ng/mL.
  Other Names: Sandimmun Neoral
  Arms: Ciclosporin
Drug: Tacrolimus — Conversion from ciclosporin to tacrolimus at target trough levels of 5-8 ng/mL in combination with/without mycophenolate mofetil and with/without steroids.
  Other Names: Prograf
  Arms: Tacrolimus

SUMMARY:
The aim of the study is to determine if the conversion from the immunosuppressive agent cyclosporine to tacrolimus contributes to an improvement of the cardiovascular risk factors, better kidney function and immune system.

DETAILED DESCRIPTION:
In addition to hypertension, diabetes, hyperlipidemia and smoking, as well as other non-traditional risk factors such as elevated C-reactive protein, homocysteine, Lp(a), or reduced renal function, depletion of endothelial progenitor cells (EPC) in the peripheral circulation may represent another important explanation for the excess cardiovascular morbidity of kidney transplant recipients. In this context, the potential association of immunosuppressive therapy with EPCs in kidney transplant recipients deserves special consideration. The use of tacrolimus associated with a more favorable cardiovascular risk factors profile in terms of improved blood pressure and lipid levels in kidney transplant recipients compared to cyclosporine users. Therefore, one can speculate whether tacrolimus users might have greater EPC counts compared to patients treated with cyclosporine.

In a pilot study we cross-sectionally studied EPC counts in 90 stable, middle-aged kidney transplant recipients. From multivariate analyses, we found a independent inverse association between EPC counts and body mass index and systolic blood pressure. Statin use was associated with greater EPC counts, while patients receiving azathioprine had lower EPC counts. These findings raised the hypothesis whether EPCs are responsible, at least in part, for the well-established association between these factors and cardiovascular outcomes.

Cystatin C is superior to serum creatinine as a marker of kidney function since cystatin C is a more sensitive marker than serum creatine for small changes in glomerular filtration rate. Until now, there are no available data on the change of cystatin C as a measure of graft function after conversion of a cyclosporine based immunosuppressive regimen to tacrolimus.

There is accumulating evidence for an important pathogenetic role of donor-reactive antibodies in kidney allograft rejection. Recent studies suggest an anti-humoral activity of tacrolimus in the setting of chronic rejection. Recent findings suggest that in patients who are on cyclosporine, tacrolimus rescue therapy could efficiently inhibit antibody formation.

Objective 1: To evaluate the change in endothelial progenitor cell (EPC) count in kidney graft recipients converted from cyclosporine to tacrolimus.

Objective 2: To evaluate the change in cystatin C as a measure of renal function in kidney graft recipients converted from cyclosporine to tacrolimus.

Objective 3: To determine the effect of tacrolimus on humoral alloreactivity in kidney graft recipients Study design: A 2:1 randomized, parallel group, open-label, prospective trial comparing two different immunosuppressive regimens in approximately 148 patients. Group A: Convert to tacrolimus in combination with/without mycophenolate mofetil and/or steroids. Group B: Maintain cyclosporine in combination with/without mycophenolate mofetil and/or steroids. Patients will be followed up for 24 months after conversion.

In an amendment (August 2006) we registered pharmacogenetic analyses of the multi-drug resistance transporter 1 (MDR1) gene (gene symbol: ABCB1). The patients´ DNA is extracted from peripheral venous blood manually with industrial extraction kits. Two gene sections are amplified by polymerase chain reaction (PCR). Mutations are determined by restriction enzymes (restriction fragment length polymorphisms, RFLP).

ELIGIBILITY:
Inclusion Criteria:

* Patient is recipient of a deceased or living donor renal transplant (including retransplants) Patient is 18 years or age or older at the time of transplantation. Patient is at least 6 months post-transplant. Patient is on a cyclosporine-based immunosuppression regimen o combination with/without mycophenolate mofetil and/or steroids at study entry.

Patient has a functioning renal allograft and estimated GFR≥39 mL/min/1.73m2 within four weeks prior to study entry.

Patient has a stable graft function without biopsy proven acute rejection episode within 3 months prior to study entry.

Patient has not experienced a cardiovascular event. Patient has fully been informed and has given written informed consent according to the International Conference on Harmonization, Good Clinical Practice.

Females are not pregnant and agree to practice effective birth control while receiving immunosuppressant medication.

Patient has indications for conversion at the investigators discretion or is suffering from cyclosporine associated side effects like hypertension, hyperlipidemia or cosmetic side effects.

Exclusion Criteria:

* Patient is recipient of a solid organ transplant other than the kidney. Patient has recurrence of primary renal disease, or de novo renal disease. Patient is pregnant or lactating. Patient had known or suspected malignancy (except for treated squamous and basal cell skin cancers) <5 years before study entry or a history of post-transplant lymphoproliferative disease (PTLD).

Patient has known hypersensitivity to tacrolimus, or any of the recipients of the drug.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2004-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Change in endothelial progenitor cells from baseline to month 24 | Baseline and 24 months
  The primary endpoint was the effect of conversion from ciclosporin to tacrolimus based immunosuppressive therapy on endothelial progenitor cell count at month 24.

SECONDARY OUTCOMES:
Renal function at baseline and after 24 months | Baseline, 24 months
  Changes in risk factors for cardiovascular outcomes like serum lipids, blood pressure, diabetes mellitus, serum C-reactive protein, body mass index. Safety was addressed according to the incidence of medical necessity to change immunosuppressive therapy, serious opportunistic infection, new-onset diabetes mellitus, cardiovascular events, malignancy, lymphoma and lymphoproliferative disease, gingival hyperplasia, hypertrichosis, alopecia, graft loss and death.

CONTACTS AND LOCATIONS:
Overall Officials: Gere Sunder-Plassmann, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Plischke M, Riegersperger M, Dunkler D, Heinze G, Kikic Z, Winkelmayer WC, Sunder-Plassmann G. Late Conversion of Kidney Transplant Recipients from Ciclosporin to Tacrolimus Improves Graft Function: Results from a Randomized Controlled Trial. PLoS One. 2015 Aug 13;10(8):e0135674. doi: 10.1371/journal.pone.0135674. eCollection 2015. PMID 26270340
- [Derived] Riegersperger M, Plischke M, Steiner S, Seidinger D, Sengoelge G, Winkelmayer WC, Sunder-Plassmann G. Effect of conversion from ciclosporin to tacrolimus on endothelial progenitor cells in stable long-term kidney transplant recipients. Transplantation. 2013 Jun 15;95(11):1338-45. doi: 10.1097/TP.0b013e31828fabb3. PMID 23594858
- See also: Website of the Medical University Vienna — http://www.meduniwien.ac.at/homepage/service/vienna-general-hospital-akh/en